CLINICAL TRIAL: NCT01695642
Title: Long-term Outcomes After Laser in Situ Keratomileusis (LASIK): Mechanical Microkeratome vs Femtosecond Laser
Brief Title: Long-term LASIK Follow up Study
Acronym: LASIK
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Roni Shtein, Assistant Professor of Ophthalmology and Visual Sciences, University of Michigan
Other Study IDs: LASIK_00049051
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Lasik Eye Surgery
Keywords: lasik, intralase, microkeratome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Microkeratome: mechanical microkeratome
- Intralase: femtosecond laser

SUMMARY:
Laser in situ keratomileusis (LASIK) is the most common corneal refractive surgery performed for correction of myopia. There are very few studies that have been performed to evaluate long-term outcomes after LASIK.

In this study, we will assess long-term outcomes 5 - 10 years after LASIK to assess stability of visual outcomes and long-term effect on corneal morphology with in vivo confocal microscopy. Clinical and corneal morphology outcomes will also be compared between patients who had flaps created with the microkeratome and femtosecond laser.

DETAILED DESCRIPTION:
Volunteers will be eligible for enrollment into the study if have had LASIK surgery for correction of myopia or myopic astigmatism at the Kellogg Eye Center with either the microkeratome or femtosecond laser for LASIK flap creation between 5 and 10 years prior.

A complete ophthalmic examination and corneal confocal microscopy will be performed. The study visit will take approximately one hour.

ELIGIBILITY:
Inclusion Criteria:

* lasik surgery at the kellogg eye center between 2002 and 2005; at least 3 months of follow up after surgery

Exclusion Criteria:

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who had LASIK surgery for correction of myopia or myopic astigmatism at the Kellogg Eye Center with either the microkeratome or femtosecond laser for LASIK flap creation between 2002 to 2005.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Compare flap creation with mikrokeratome and Intralase | 8 to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Roni Shtein, MD, MS, Principal Investigator — University of Michigan Kellogg Eye Center
Locations (1):
- Kellogg Eye Center, Ann Arbor, Michigan, United States